CLINICAL TRIAL: NCT03990519
Title: A Randomized, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of a Single Subcutaneous Dose of JNJ-26366821 in Healthy Volunteers
Brief Title: A Study of a Single Subcutaneous Dose of JNJ-26366821 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108637; 26366821RSS1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — RWJ 800088

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort1: JNJ-2636682/Placebo (Experimental): Participants will receive single dose of JNJ-26366821 or placebo on Day 1.
  Interventions: Drug: JNJ-26366821; Drug: Placebo
- Cohort 2: JNJ-26366821/Placebo (Experimental): Participants will receive single dose of JNJ-26366821 or placebo on Day 1.
  Interventions: Drug: JNJ-26366821; Drug: Placebo
- Cohort 3: JNJ-26366821/Placebo (Experimental): Participants will receive single dose of JNJ-26366821 or placebo. The dose of JNJ-26366821 will be selected based on the safety, pharmacodynamics, and pharmacokinetics data from the previous Cohorts 1 and 2.
  Interventions: Drug: JNJ-26366821; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-26366821 — Participants will receive sterile solution of JNJ-26366821 subcutaneously (SC).
Drug: Placebo — Participants will receive sodium chloride injection as placebo on Day 1.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single subcutaneous (SC) dose of JNJ-26366821.

ELIGIBILITY:
Inclusion Criteria:

* Overall good health, on the basis of full physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Body weight 50 - 100 kilogram (kg), body mass index (BMI) 18 - 30 kilogram per meter square (kg/m^2), inclusive at screening
* Platelet count within range: 145 to 350*10^9/liter (L), inclusive at screening
* Hematologic values, coagulation profile, renal and liver function within normal range at screening or if out of range and considered not clinically significant by the investigator
* Non-smoker for at least the previous 3 months prior to screening and negative urine cotinine test at screening and admission

Exclusion Criteria:

* History of any clinically significant medical illness or disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Has a disease or disease treatment history associated with immune suppression or lymphopenia, these include but are not limited to bone marrow or organ transplantation, lymphoproliferative disorders, T- or B-cell deficiency syndromes, splenectomy, functional asplenism, and chronic granulomatous disease
* Has a personal history of genetic or congenital prothrombotic condition or new conditions associated with thromboembolic events or bleeding disorders, including (but not limited to) myocardial infarction, cerebral vascular accident/stroke, deep vein thrombosis, pulmonary embolism, hemophilia, or menometrorrhagia
* Participants who had received hematopoietic growth factors within 3 months prior to study drug administration
* Donation of blood or blood components within 90 days prior to drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) as a Measure of Safety and Tolerability | Up to Day 30
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-26366821 | Day 1: predose, 1, 4, 12 hours (hrs) postdose; Day 2: 24 and 36 hrs postdose; Day 3: 48 and 60 hrs postdose; Day 4: 72 hrs postdose; Day 5: 96 hrs; Day 6: 120 hrs postdose; Days 15 and 30
  Cmax is defined as the maximum observed plasma concentration of JNJ- 26366821.
Area Under the Plasma Concentration Versus Time Curve from Time 0 to Time of the Last Measurable Concentration AUC0-Last of JNJ-26366821 | Day 1: predose, 1, 4, 12 hours (hrs) postdose; Day 2: 24 and 36 hrs postdose; Day 3: 48 and 60 hrs postdose; Day 4: 72 hrs postdose; Day 5: 96 hrs; Day 6: 120 hrs postdose; Days 15 and 30
  AUC 0-last is defined as area under the plasma concentration versus time curve from time 0 to time of the last measurable concentration of JNJ-26366821 will be assessed.
Apparent Elimination Half-Life (t1/2) of JNJ-26366821 | Day 1: predose, 1, 4, 12 hours (hrs) postdose; Day 2: 24 and 36 hrs postdose; Day 3: 48 and 60 hrs postdose; Day 4: 72 hrs postdose; Day 5: 96 hrs; Day 6: 120 hrs postdose; Days 15 and 30
  T1/2 is define as apparent elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve.
Area Under the JNJ-26366821 Concentration Versus Time Curve from Time 0 to Infinite Time (AUC[0-infinity]) of JNJ-26366821 | Day 1: predose, 1, 4, 12 hours (hrs) postdose; Day 2: 24 and 36 hrs postdose; Day 3: 48 and 60 hrs postdose; Day 4: 72 hrs postdose; Day 5: 96 hrs; Day 6: 120 hrs postdose; Days 15 and 30
  AUC (0-infinity) is defined as area under the JNJ-26366821 concentration Versus time curve from Time 0 to infinite time.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-26366821 | Day 1: predose, 1, 4, 12 hours (hrs) postdose; Day 2: 24 and 36 hrs postdose; Day 3: 48 and 60 hrs postdose; Day 4: 72 hrs postdose; Day 5: 96 hrs; Day 6: 120 hrs postdose; Days 15 and 30
  Tmax is defined as time to reach the maximum observed plasma JNJ-26366821 concentration.
Change in Platelet Count from Baseline at Each Dose and Time | Baseline up to Day 30
  Change from baseline in platelet count at each dose and time will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Harbor Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency